CLINICAL TRIAL: NCT03748563
Title: Accuracy of Magnetically Maneuvered Capsule Endoscopy for Detection of Esophagogastric Varices in Patients With Cirrhosis
Brief Title: Accuracy of Magnetically Maneuvered Capsule Endoscopy for Detection of EGV in Patients With Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Ruijin Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Shanghai East Hospital of Tongji University (Other); Yangpu District Central Hospital Affiliated to Tongji University (Other); Zhujiang Hospital (Other); Qilu Hospital of Shandong University (Other); The Third Xiangya Hospital of Central South University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The Fifth Affiliated Hospital of Zunyi Medical College (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Shanghai Pudong New Area Gongli Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Professor, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CENTERS
Record Dates: First submitted 2018-11-12; First posted 2018-11-21 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Liver Cirrhosis; Portal Hypertension; Esophageal Varices; Gastric Varix
Keywords: Capsule Endoscopy; Liver Cirrhosis; Esophageal Varices; Gastric Varices; Portal hypertensive gastropathy; Portal hypertensive enteropathy
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal; Esophageal and Gastric Varices | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Intervention Model Description: Diagnostic accuracy study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ds-MCE and EGD (Experimental): All the enrolled participants will undergo the examination of detachable string magnetically maneuvered capsule endoscopy (ds-MCE) first, followed by EGD within 48 hours.
  Interventions: Diagnostic Test: ds-MCE and EGD

INTERVENTIONS:
Diagnostic Test: ds-MCE and EGD — Procedure of ds-MCE:
  The ds-MCE system mainly consists of two parts: the NaviCam magnetically maneuvered capsule endoscopy system and the detachable string part. The capsule, which is partially enclosed within the sleeve, can be actively moved in the esophagus through the control of string. Investigator can examine the entire esophagus several times under real time views. After completing the esophageal examination, the capsule could be detached from the string through injecting air into the hollow string with the syringe. Then, the examination of stomach under magnetic control and small bowel under the natural action of gastrointestinal peristalsis follows.
  Procedure of EGD:
  The esophagogastroduodenoscopy (EGD) will be performed using conventional upper gastrointestinal video endoscopy, according to the standard procedure at individual centers. EGD will be performed within 48 hours after ds-MCE procedure and usually during the same endoscopic session.

SUMMARY:
This is a diagnostic accuracy study. Eligible individuals will be enrolled and asked to undergo ds-MCE and EGD examinations. EGD is the reference standard against which ds-MCE is compared, and it will be performed within 48 hours after ds-MCE examination. The primary outcome is the sensitivity and specificity of ds-MCE in identifying the presence of esophagogastric (EGV) in patients with cirrhosis, using detection by EGD as the reference. The diagnostic accuracy of ds-MCE in detection of high-risk EV, high-risk EGV, EV, large EV, red signs of EV, GV, cardiofundal GV and PHG compared with the EGD will also be assessed. The incidence of PHE in small bowel under ds-MCE, the examination time of ds-MCE and EGD procedures, patient satisfaction assessment and safety evaluation will also be evaluated.

DETAILED DESCRIPTION:
Cirrhosis is the major cause of liver disease-related morbidity and mortality worldwide. Portal hypertension (PH) is the hemodynamic abnormality in patients with cirrhosis, which is associated with various pathological changes throughout the entire gastrointestinal tract, manifesting as esophagogastric varices (EGV), portal hypertensive gastropathy (PHG), and portal hypertensive enteropathy (PHE). Baveno consensus and other practice guidelines recommended that patients with cirrhosis undergo endoscopic screening for EGV at the time of diagnosis and undergo periodic surveillance endoscopy throughout the whole course of cirrhosis.

Esophagogastroduodenoscopy (EGD) is recognized as the gold standard for detection and follow-up of EGV in cirrhotic patients, allowing for direct mucosal visualization and therapeutic intervention. EGD is however an invasive procedure and there is potential for procedure-related complications, such as perforation and bleeding. Besides, conscious sedation is always required, leading to increased cost, risk, and inconvenience for the patients.These factors lead to a decrease of patient compliance as well as the effectiveness of the screening program.

The capsule endoscopy (CE) system provides a noninvasive and relatively comfortable approach to visualize the GI tract, and the development of esophageal capsule endoscopy (ECE) makes it possible to capture clear images of esophagus without the need of sedation. However, the accuracy of ECE is not currently sufficient to replace EGD for the detection and grading for the esophageal varices. Besides, previous studies presented that the sensitivity of ECE for detecting gastric varices (GVs) and PHG varies from 3% to 69%, which denoted ECE was far from a suitable alternative for diagnosing gastric lesions.

To overcome these limitations, a new technique, so-called detachable string magnetically maneuvered capsule endoscopy (ds-MCE) was developed. The ds-MCE system consists of two parts: the magnetically maneuvered capsule endoscopy (MCE) system and a transparent latex sleeve with a hollow string. One end of the hollow string is a transparent thin latex sleeve that can be wrapped on the surface of the capsule, and the other end of the string is connected to the syringe. The capsule, which is partially enclosed within the sleeve, can be actively moved in the esophagus through the control of string. In this case, investigator can examine the entire esophageal mucosa several times under real time views. The capsule then can be detached from the string system through injecting air into the hollow string with the syringe after completing the examination of esophagus. The magnetic capsule in the stomach can be accurately controlled through multidimensional rotation and adaptive matching of an external C-arm robot. Previous studies have demonstrated that the diagnostic accuracy of MCE for detecting gastric focal lesions is comparable with that of conventional EGD. Two previously studies of ds-MCE confirmed it was a feasible, safe and well-tolerated method for completely viewing esophagus and stomach, without the need for sedation. Besides, the 8-10h battery life of the ds-MCE enables complete examination of the small bowel, which enables to provide a more comprehensive evaluation of gastrointestinal changes.

Considering all these backgrounds, in the current prospective study, the primary aim is to assess the diagnostic performance of the ds-MCE in identifying the presence of EGV in cirrhotic patients, using EGD as the reference standard. The diagnostic accuracy of ds-MCE in detection of high-risk EV, high-risk EGV, EV, large EV, red signs of EV, GV, cardiofundal GV and PHG compared with the EGD will also be assessed. The incidence of PHE in small bowel under ds-MCE, the examination time of ds-MCE and EGD procedures, patient satisfaction assessment and safety evaluation will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Gender is not limited.
2. Patients aged 18 years or older.
3. Both inpatients and outpatients.
4. Clinically evident or biopsy-proven liver cirrhosis.
5. Able to provide informed consent.

Exclusion Criteria:

1. Patients aged less than 18 years.
2. Patients with Zenker's diverticulum.
3. Patients with active gastrointestinal bleeding.
4. Patients who have participated in or are participating in other clinical trials.
5. Pregnancy or suspected pregnancy.
6. Suspected or known intestinal stenosis or other known risk factors for capsule retention.
7. Pacemaker or other implanted electromedical devices which could interfere with magnetic resonance.
8. Patients with dysphagia.
9. Life-threatening conditions.
10. Patients plan to undergo magnetic resonance imaging examination before excretion of the MCE.
11. Patients who refuse to give informed consent.
12. Patients with any condition that precludes compliance with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
the diagnostic accuracy of the ds-MCE in identifying the presence of esophagogastric varices (EGV) | 2 weeks
  the sensitivity and specificity of ds-MCE in identifying EGV in patients with cirrhosis, using the detection by EGD as the reference.

SECONDARY OUTCOMES:
the diagnostic accuracy of the ds-MCE in identifying the presence of esophageal varices (EV) | 2 weeks
  The sensitivity, specificity, PPV, NPV and overall diagnostic accuracy of ds-MCE in detection of EV, using the detection by EGD as the reference.
the diagnostic accuracy of the ds-MCE in identifying the red sign of EV | 2 weeks
  The sensitivity, specificity, PPV, NPV and overall diagnostic accuracy of ds-MCE in identifying the red sign of EV, using the detection by EGD as the reference.
the diagnostic accuracy of the ds-MCE in differentiating large esophageal varices | 2 weeks
  The sensitivity, specificity, PPV, NPV and overall diagnostic accuracy of ds-MCE in detection of large EV, using the detection by EGD as the reference.
the optimal esophageal luminal circumference percentage threshold under ds-MCE for distinguishing large EV | 2 weeks
  To investigate the optimal threshold of the proportion of ds-MCE esophageal luminal circumference occupied by the largest esophageal varix present in differentiating large EV from small or no EV, using the detection by EGD as the reference.
the diagnostic accuracy of the ds-MCE in differentiating high-risk esophageal varices | 2 weeks
  The sensitivity, specificity, PPV, NPV and overall diagnostic accuracy of ds-MCE in detection of high-risk EV, using the detection by EGD as the reference.
the diagnostic accuracy of the ds-MCE in detection of high-risk EGV | 2 weeks
  The sensitivity, specificity, PPV, NPV and overall diagnostic accuracy of ds-MCE in detection of high-risk EGV, using the detection by EGD as the reference.
the diagnostic accuracy of the ds-MCE in detecting gastric varices (GV) | 2 weeks
  The sensitivity, specificity, PPV, NPV and overall diagnostic accuracy of ds-MCE in detection of GV, using the detection by EGD as the reference.
the diagnostic accuracy of the ds-MCE in detecting cardiofundal gastric varices | 2 weeks
  The sensitivity, specificity, PPV, NPV and overall diagnostic accuracy of ds-MCE in detection of cardiofundal GV, using the detection by EGD as the reference.
the diagnostic accuracy of the ds-MCE in identifying portal hypertensive gastropathy | 2 weeks
  The sensitivity, specificity, PPV, NPV and overall diagnostic accuracy of ds-MCE in detection of portal hypertensive gastropathy (PHG), using the detection by EGD as the reference.
the incidence of portal hypertensive enteropathy (PHE) under ds-MCE | 2 weeks
  Endoscopic findings of PHE include mucosal inflammatory-like abnormalities, vascular lesions and spontaneous bleeding.
the examination time of ds-MCE and EGD | 2 weeks
  Examination time of ds-MCE include esophageal transit time (ETT), gastric examination time (GET), gastric transit time (GTT), small bowel transit time (SBTT), and total running time (TRT). Examination time of EGD is the time from the endoscope entering to exiting from the esophagus.
patient satisfaction evaluation of the ds-MCE and EGD | 2 weeks
  Patient satisfaction score of ds-MCE and EGD procedures.
Safety evaluation | 2 weeks
  All adverse events occurring during the study will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, Principal Investigator — Changhai Hospital
Locations (14):
- China (14):
  - Zhujiang Hospital,Southern Medical University, Guangzhou, Guangdong
  - the Fifth Affiliated Hospital of Zunyi Medical University, Zhuhai, Guangdong
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Jiao Tong University affiliated Sixth people's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tongji Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Pudong New Area Gongli Hospital, Shanghai, Shanghai Municipality
  - Yangpu District Central Hospital Affiliated to Tongji University, Shanghai, Shanghai Municipality
  - First Affiliated Hospital Xi'an Jiaotong University, Xi’an, Shanxi
  - The First Affiliated Hospital of Zhejiang Chinese Medical University, Hanzhou, Zhejiang
  - Changhai Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared after publication of the main results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years.
Access Criteria: The website of the journal where the results published, and ClinicalTrials.gov web site.

REFERENCES:
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] North Italian Endoscopic Club for the Study and Treatment of Esophageal Varices. Prediction of the first variceal hemorrhage in patients with cirrhosis of the liver and esophageal varices. A prospective multicenter study. N Engl J Med. 1988 Oct 13;319(15):983-9. doi: 10.1056/NEJM198810133191505. PMID 3262200
- [Background] Spina GP, Arcidiacono R, Bosch J, Pagliaro L, Burroughs AK, Santambrogio R, Rossi A. Gastric endoscopic features in portal hypertension: final report of a consensus conference, Milan, Italy, September 19, 1992. J Hepatol. 1994 Sep;21(3):461-7. doi: 10.1016/s0168-8278(05)80329-0. No abstract available. PMID 7836719
- [Background] Sarin SK, Lahoti D, Saxena SP, Murthy NS, Makwana UK. Prevalence, classification and natural history of gastric varices: a long-term follow-up study in 568 portal hypertension patients. Hepatology. 1992 Dec;16(6):1343-9. doi: 10.1002/hep.1840160607. PMID 1446890
- [Background] Kodama M, Uto H, Numata M, Hori T, Murayama T, Sasaki F, Tsubouchi N, Ido A, Shimoda K, Tsubouchi H. Endoscopic characterization of the small bowel in patients with portal hypertension evaluated by double balloon endoscopy. J Gastroenterol. 2008;43(8):589-96. doi: 10.1007/s00535-008-2198-1. Epub 2008 Aug 17. PMID 18709480
- [Background] D'Amico G, De Franchis R; Cooperative Study Group. Upper digestive bleeding in cirrhosis. Post-therapeutic outcome and prognostic indicators. Hepatology. 2003 Sep;38(3):599-612. doi: 10.1053/jhep.2003.50385. PMID 12939586
- [Background] Garcia-Tsao G, Sanyal AJ, Grace ND, Carey W; Practice Guidelines Committee of the American Association for the Study of Liver Diseases; Practice Parameters Committee of the American College of Gastroenterology. Prevention and management of gastroesophageal varices and variceal hemorrhage in cirrhosis. Hepatology. 2007 Sep;46(3):922-38. doi: 10.1002/hep.21907. No abstract available. PMID 17879356
- [Background] Lapalus MG, Dumortier J, Fumex F, Roman S, Lot M, Prost B, Mion F, Ponchon T. Esophageal capsule endoscopy versus esophagogastroduodenoscopy for evaluating portal hypertension: a prospective comparative study of performance and tolerance. Endoscopy. 2006 Jan;38(1):36-41. doi: 10.1055/s-2006-924975. PMID 16429353
- [Background] Gralnek IM, Adler SN, Yassin K, Koslowsky B, Metzger Y, Eliakim R. Detecting esophageal disease with second-generation capsule endoscopy: initial evaluation of the PillCam ESO 2. Endoscopy. 2008 Apr;40(4):275-9. doi: 10.1055/s-2007-995645. PMID 18389444
- [Background] de Franchis R, Eisen GM, Laine L, Fernandez-Urien I, Herrerias JM, Brown RD, Fisher L, Vargas HE, Vargo J, Thompson J, Eliakim R. Esophageal capsule endoscopy for screening and surveillance of esophageal varices in patients with portal hypertension. Hepatology. 2008 May;47(5):1595-603. doi: 10.1002/hep.22227. PMID 18435461
- [Derived] Jiang X, Pan J, Xu Q, Song YH, Sun HH, Peng C, Qi XL, Qian YY, Zou WB, Yang Y, Jin SQ, Duan BS, Wu S, Chu Y, Xiao DH, Hu LJ, Cao JZ, Dai JF, Liu X, Xia T, Zhou W, Chen T, Zhou CH, Wu W, Liu SJ, Yang ZY, Wang F, Zhang L, Li CZ, Xu H, Wang JX, Wei B, Lin Y, Deng X, Qu LH, Shen YQ, Wang H, Huang YF, Bao HB, Zhang S, Li L, Shi YH, Wang XY, Zou DW, Wan XJ, Xu MD, Mao H, He CH, Li Z, Zuo XL, He SX, Xie XP, Liu J, Yang CQ, Spada C, Li ZS, Liao Z. Diagnostic accuracy of magnetically guided capsule endoscopy with a detachable string for detecting oesophagogastric varices in adults with cirrhosis: prospective multicentre study. BMJ. 2024 Mar 5;384:e078581. doi: 10.1136/bmj-2023-078581. PMID 38443074

DOCUMENTS (2):
  • Study Protocol (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT03748563/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT03748563/SAP_001.pdf